CLINICAL TRIAL: NCT01001169
Title: Safety and Immunogenicity Study of GSK Biologicals' Pandemic Influenza (H1N1) Candidate Vaccine (GSK2340274A) in Japanese Children Aged 6 Months to 17 Years
Brief Title: Safety and Immunogenocity Study of GSK Biologicals' Pandemic Influenza (H1N1) Candidate Vaccine in Japanese Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 113847
Record Dates: First submitted 2009-10-22; First posted 2009-10-23 (Estimated); Results first posted 2017-05-02 (Actual); Last update posted 2018-08-17 (Actual); Status verified 2018-07

CONDITIONS: Influenza
Keywords: GSK Bio's influenza vaccine GSK2340274A; influenza infection
MeSH Terms: conditions — Influenza, Human

ARMS (2):
- GSK2340274A_F1 6M-9Y GROUP (Experimental): Healthy male or female Japanese children, between and including 6 months to 9 years of age, who received two doses of GSK2340274A vaccine (formulation 1), administered intramuscularly into the deltoid region of the arm (intramuscularly into the anterolateral part of the thigh for subjects below 12 months of age at the entry of the study), according to 0, 21-day schedule. Within this group, enrolment of subjects was stratified by age into two subgroups, from 6 to 35 months and from 3 to 9 years.
  Interventions: Biological: GSK Biologicals' Pandemic influenza (H1N1) candidate vaccine (GSK2340274A)
- GSK2340274A_F2 10Y-17Y GROUP (Experimental): Healthy male or female Japanese children, between and including 10 to 17 years of age, who received two doses of GSK2340274A vaccine (formulation 2), administered intramuscularly into the deltoid region of the arm, according to 0, 21-day schedule.
  Interventions: Biological: GSK Biologicals' Pandemic influenza (H1N1) candidate vaccine (GSK2340274A)

INTERVENTIONS:
Biological: GSK Biologicals' Pandemic influenza (H1N1) candidate vaccine (GSK2340274A) — Two intramuscular injections

SUMMARY:
The objective of this study is to evaluate the immunogenicity and safety of GSK Biologicals' investigational influenza vaccine GSK2340274A following one dose and following a second dose, using the same dosage as has been used in the H5N1 development program in Japanese children aged 10-17 years and an alternative dose in children aged 6 months to 9 years.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that their parent(s)/Legally Acceptable Representative(s) (LAR) can and will comply with the requirements of the protocol.
* Japanese children, male or female, aged between 6 months and 17 years at the time of the first study vaccination.
* Written informed consent obtained from the subject's parent(s) or LAR(s) of the subject. Whenever possible, an assent should also be obtained from the subject.
* Healthy children as established by medical history and clinical examination when entering into the study (Particular attention must be exercised when dealing with patients with bronchial asthma).
* Parent/LAR with access to a consistent means of telephone contact, land line or mobile, but NOT a pay phone or other multiple-user device.
* Female subjects of childbearing potential may be enrolled in the study, if the subject: has practiced adequate contraception for 30 days prior to vaccination, and has a negative pregnancy test on the day of vaccination, and has agreed to continue adequate contraception during the entire treatment period and for 2 months after completion of the vaccination series.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine within 30 days preceding the first dose of the study vaccine or planned use during the study period.
* Clinically or virologically confirmed influenza infection from May 2009 to the day of enrolment.
* Previous administration of a novel [H1N1]v vaccine.
* Administration of any vaccines within 30 days before vaccination or planned administration within the first vaccination up to blood sampling at Day 42 and within 30 days prior to blood sampling at Day 182, with the exception of seasonal influenza vaccine.
* Administration of any seasonal influenza vaccine within 14 days before vaccination on Day 0, or planned administration within the first vaccination up to blood sampling at Day 42 and within 14 days prior to blood sampling at Day 182.
* Excessive underweight or excessive obesity. (Under or upper 2-fold standard deviation of weight distribution that are corresponding age group are used as reference).
* Chronic administration of immunosuppressants or other immune-modifying drugs within three months prior to enrolment in this study or planned administration during the study period.
* Acute disease and/or fever at the time of enrolment:
* Fever is defined as temperature >= 37.5°C on oral, axillary or tympanic setting, or >= 38.0°C on rectal setting.
* Subjects with a minor illness (such as mild diarrhoea, mild upper respiratory infection) without fever may be enrolled at the discretion of the investigator.
* Any confirmed or suspected immunosuppressive or immunodeficient condition based on medical history and physical examination (no laboratory testing required).
* Acute or chronic, clinically-significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by medical history and physical examination.
* Administration of immunoglobulins and/or any blood products within the three months prior to the enrolment in this study, or planned during the study.
* Any known or suspected allergy to any constituent of influenza vaccines; a history of anaphylactic-type reaction to consumption of eggs; or a history of severe adverse reaction to a previous influenza vaccine.
* History of any neurological disorder including acute disseminated encephalomyelitis and Guillain-Barré syndrome, or convulsive seizures and epilepsy.
* Any significant disorder of coagulation or treatment with warfarin derivatives or heparin. Persons receiving individual doses of low molecular weight heparin are eligible if no such doses are given in the 24 hours before a study vaccination. Persons receiving prophylactic antiplatelet medications, e.g., low-dose acetylsalicylic acid, and without a clinically-apparent bleeding tendency, are eligible
* Any conditions which, in the opinion of the investigator, prevents the subject from participating to the study.
* Child in Care.

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2009-10-01; Primary Completion 2010-05-17 (Actual); Study Completion 2010-05-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Van Damme P, Kafeja F, Bambure V, Hanon E, Moris P, Roman F, Gillard P. Long-term persistence of humoral and cellular immune responses induced by an AS03A-adjuvanted H1N1 2009 influenza vaccine: an open-label, randomized study in adults aged 18-60 years and older. Hum Vaccin Immunother. 2013 Jul;9(7):1512-22. doi: 10.4161/hv.24504. Epub 2013 Apr 9. PMID 23571166
- [Derived] Saitoh A, Nagai A, Tenjinbaru K, Li P, Vaughn DW, Roman F, Kato T. Safety and persistence of immunological response 6 months after intramuscular vaccination with an AS03-adjuvanted H1N1 2009 influenza vaccine: an open-label, randomized trial in Japanese children aged 6 months to 17 years. Hum Vaccin Immunother. 2012 Jun;8(6):749-58. doi: 10.4161/hv.19684. Epub 2012 Apr 12. PMID 22495117
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 113847 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 113847 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 113847 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 113847 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 113847 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 113847 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 113847 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | GSK2340274A_F1 6M-9Y Group | GSK2340274A_F2 10Y-17Y Group
Started | 30 | 30
Completed | 28 | 29
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK2340274A_F1 6M-9Y Group | GSK2340274A_F2 10Y-17Y Group | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: Months] | 49.00 (27.66) | 163.00 (32.41) | 106.00 (64.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 18 | 34
  Male | 14 | 12 | 26

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Haemagglutination Inhibition (HI) Antibody Concentrations Above the Cut-off Value
Description: The cut-off values for the humoral immune response in terms of vaccine H1N1 HI antibodies were equal to or above (≥) 1:10.
  The Flu strain assessed was A/California/7/2009 (H1N1)v-like virus (Flu A/CAL/7/09), in subjects aged between 6 months to 9 years and 10 to 17 years, following the Committee for Medicinal Products for Human Use (CHMP) and the Center for Biologics Evaluation and Research (CBER) guidance.
Time Frame: At Day 42
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity at Day 42, which included all evaluable subjects for whom assay results for antibodies against A/California-like HA antigen for the blood samples taken on Day 42 (21 days after the second vaccination) were available.
Measure: Number; unit: Subjects
Arm/Group | GSK2340274A_F1 6M-9Y Group | GSK2340274A_F2 10Y-17Y Group
Number analyzed (Participants) | 28 | 30
Subjects | 28 | 30

2. Primary Outcome: Titers for Serum HI Antibodies Against Flu A/CAL/7/09 Strain of Influenza Disease
Description: Titers are presented as geometric mean titers (GMTs). The reference seropositivity cut-off value was ≥ 1:10. The Flu strain assessed was Flu A/CAL/7/09, in subjects aged between 6 months to 9 years and 10 to 17 years, following the CHMP and the CBER guidance.
Time Frame: At Day 42
Population: The analysis was performed on the ATP cohort for immunogenicity at Day 42, which included all evaluable for whom assay results for antibodies against A/California-like HA antigen for the blood samples taken on Day 42 (21 days after the second vaccination) were available.
Measure: Geometric Mean (97.5% Confidence Interval); unit: Titers
Arm/Group | GSK2340274A_F1 6M-9Y Group | GSK2340274A_F2 10Y-17Y Group
Number analyzed (Participants) | 28 | 30
Titers | 939.3 [722.9 to 1220.6] | 874.3 [717.4 to 1065.4]

3. Primary Outcome: Number of Seroconverted Subjects for HI Antibodies
Description: Seroconversion (SCR) was defined as follows:
  For initially seronegative subjects, antibody titer ≥ 1:40 after vaccination; For initially seropositive subjects, antibody titer after vaccination ≥ 4 fold the pre-vaccination antibody titer. The Flu strain assessed was Flu A/CAL/7/09, in subjects aged between 6 months to 9 years and 10 to 17 years, following the CHMP and the CBER guidance.
  The CBER criterion was fulfilled if the lower 97.5% confidence interval for SCR was > 40%.
  The CHMP criterion was fulfilled if the point estimate for SCR was > 40%.
Time Frame: At Day 42
Population: as for outcome 2
Measure: Number; unit: Subjects
Arm/Group | GSK2340274A_F1 6M-9Y Group | GSK2340274A_F2 10Y-17Y Group
Number analyzed (Participants) | 28 | 30
Subjects | 28 | 30

4. Primary Outcome: Number of Seroprotected Subjects for HI Antibodies
Description: A seroprotected subject was defined as a vaccinated subject with a serum hemagglutination inhibition (HI) titer equal to or above (≥) 1:40. The Flu strain assessed was Flu A/CAL/7/09, in subjects aged between 6 months to 9 years and 10 to 17 years, following the CHMP and the CBER guidance.
  The CBER Criterion was fulfilled if the lower 97.5% confidence interval for seroprotection (SPR) was > 70%.
  The CHMP Criterion was fulfilled if the post-vaccination point estimate for SPR was > 70%.
Time Frame: At Day 42
Population: as for outcome 2
Measure: Number; unit: Subjects
Arm/Group | GSK2340274A_F1 6M-9Y Group | GSK2340274A_F2 10Y-17Y Group
Number analyzed (Participants) | 28 | 30
Subjects | 28 | 30

5. Primary Outcome: Geometric Mean Fold Rise (GMFR) for HI Antibodies Against Flu A/CAL/7/09 Strain of Influenza Disease
Description: GMFR, also called seroconversion factor (SCF), was defined as the fold increase in serum HI GMTs post-vaccination compared to pre-vaccination. The Flu strain assessed was Flu A/CAL/7/09, in subjects aged between 6 months to 9 years and 10 to 17 years, following the CHMP guidance.
  The CHMP Criterion was fulfilled if the point estimate for GMFR was > 2.5.
Time Frame: At Day 42
Population: as for outcome 2
Measure: Geometric Mean (97.5% Confidence Interval); unit: Titers
Arm/Group | GSK2340274A_F1 6M-9Y Group | GSK2340274A_F2 10Y-17Y Group
Number analyzed (Participants) | 28 | 30
Titers | 146.8 [99.6 to 216.4] | 57.1 [33.5 to 97.3]

6. Secondary Outcome: Number of Subjects With HI Antibody Concentrations Above the Cut-off Value
Description: The cut-off values for the humoral immune response in terms of vaccine H1N1 HI antibodies were equal to or above (≥) 1:10. The Flu strain assessed was Flu A/CAL/7/09, in subjects aged between 6 months to 9 years and 10 to 17 years, following the CHMP and the CBER guidance.
Time Frame: At Days 0 and 21
Population: The analysis was performed on the ATP cohort for immunogenicity at Day 21, which included all evaluable for whom assay results for antibodies against A/California-like HA antigen for the blood sample taken 21 days after the first vaccination were available.
Measure: Number; unit: Subjects
Groups:
- GSK2340274A_F1 6M-35M Subgroup: Healthy male or female Japanese children, between and including 6 to 35 months of age, who received two doses of GSK2340274A vaccine (formulation 1), administered intramuscularly into the deltoid region of the arm (intramuscularly into the anterolateral part of the thigh for subjects below 12 months of age at the entry of the study), according to 0, 21-day schedule.
- GSK2340274A_F1 3Y-9Y Subgroup: Healthy male or female Japanese children, between and including 3 to 9 years of age, who received two doses of GSK2340274A vaccine (formulation 1), administered intramuscularly into the deltoid region of the arm, according to 0, 21-day schedule.
Arm/Group | GSK2340274A_F1 6M-9Y Group | GSK2340274A_F2 10Y-17Y Group | GSK2340274A_F1 6M-35M Subgroup | GSK2340274A_F1 3Y-9Y Subgroup
Number analyzed (Participants) | 29 | 30 | 10 | 19
Subjects
  Flu A/CAL/7/09, Day 0 | 5 | 18 | 0 | 5
  Flu A/CAL/7/09, Day 21 | 29 | 30 | 10 | 19

7. Secondary Outcome: Number of Subjects With HI Antibody Concentrations Above the Cut-off Value
Description: The cut-off values for the humoral immune response in terms of vaccine H1N1 HI antibodies were equal to or above (≥) 1:10. The Flu strain assessed was Flu A/CAL/7/09, in subjects aged between 6 months to 9 years, following the CHMP and the CBER guidance.
  Note: Analyses based on 95% CI for 10-17 year age category at Day 42 were not performed.
Time Frame: At Days 0 and 42
Population: as for outcome 2
Measure: Number; unit: Subjects
Arm/Group | GSK2340274A_F1 6M-35M Subgroup | GSK2340274A_F1 3Y-9Y Subgroup
Number analyzed (Participants) | 9 | 19
Subjects
  Flu A/CAL/7/09, Day 0 | 0 | 5
  Flu A/CAL/7/09, Day 42 | 9 | 19

8. Secondary Outcome: Number of Subjects With HI Antibody Concentrations Above the Cut-off Value
Description: as for outcome 6
Time Frame: At Days 0 and 182
Population: The analysis was performed on the ATP cohort for immunogenicity at Day 182, which included all evaluable subjects for whom assay results for antibodies against A/California-like HA antigen for the blood samples taken on Day 182 were available.
Measure: Number; unit: Subjects
Arm/Group | GSK2340274A_F1 6M-9Y Group | GSK2340274A_F2 10Y-17Y Group | GSK2340274A_F1 6M-35M Subgroup | GSK2340274A_F1 3Y-9Y Subgroup
Number analyzed (Participants) | 28 | 29 | 9 | 19
Subjects
  Flu A/CAL/7/09, Day 0 | 5 | 17 | 0 | 5
  Flu A/CAL/7/09, Day 182 | 28 | 29 | 9 | 19

9. Secondary Outcome: Titers for Serum HI Antibodies Against Flu A/CAL/7/09 Strain of Influenza Disease
Description: as for outcome 2
Time Frame: At Days 0 and 21
Population: The analysis was performed on the ATP cohort for immunogenicity at Day 21, which included all evaluable subjects for whom assay results for antibodies against A/California-like HA antigen for the blood sample taken 21 days after the first vaccination were available.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | GSK2340274A_F1 6M-9Y Group | GSK2340274A_F2 10Y-17Y Group | GSK2340274A_F1 6M-35M Subgroup | GSK2340274A_F1 3Y-9Y Subgroup
Number analyzed (Participants) | 29 | 30 | 10 | 19
Titers
  Flu A/CAL/7/09, Day 0 | 6.3 [5.0 to 8.1] | 15.3 [9.5 to 24.6] | NA [NA to NA] — Value below the cut-off value for the respective assay. | 7.2 [5.0 to 10.3]
  Flu A/CAL/7/09, Day 21 | 172.0 [130.1 to 227.6] | 339.0 [238.8 to 481.2] | 117.3 [72.2 to 190.8] | 210.4 [150.4 to 294.5]

10. Secondary Outcome: Titers for Serum HI Antibodies Against Flu A/CAL/7/09 Strain of Influenza Disease
Description: Titers are presented as geometric mean titers (GMTs). The reference seropositivity cut-off value was ≥ 1:10. The Flu strain assessed was Flu A/CAL/7/09, in subjects aged between 6 months to 9 years, following the CHMP and the CBER guidance.
  Note: Analyses based on 95% CI for 10-17 year age category at Day 42 were not performed.
Time Frame: At Days 0 and 42
Population: The analysis was performed on the ATP cohort for immunogenicity at Day 42, which included all evaluable subjects for whom assay results for antibodies against A/California-like HA antigen for the blood samples taken on Day 42 (21 days after the second vaccination) were available.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | GSK2340274A_F1 6M-35M Subgroup | GSK2340274A_F1 3Y-9Y Subgroup
Number analyzed (Participants) | 9 | 19
Titers
  Flu A/CAL/7/09, Day 0 | NA [NA to NA] — Value below the cut-off value for the respective assay. | 7.2 [5.0 to 10.3]
  Flu A/CAL/7/09, Day 42 | 1279.9 [806.9 to 2030.4] | 811.3 [628.4 to 1047.4]

11. Secondary Outcome: Titers for Serum HI Antibodies Against Flu A/CAL/7/09 Strain of Influenza Disease
Description: as for outcome 2
Time Frame: At Days 0 and 182
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | GSK2340274A_F1 6M-9Y Group | GSK2340274A_F2 10Y-17Y Group | GSK2340274A_F1 6M-35M Subgroup | GSK2340274A_F1 3Y-9Y Subgroup
Number analyzed (Participants) | 28 | 29 | 9 | 19
Titers
  Flu A/CAL/7/09, Day 0 | 6.4 [5.0 to 8.2] | 14.8 [9.1 to 24.1] | NA [NA to NA] — Value below the cut-off value for the respective assay. | 7.2 [5.0 to 10.3]
  Flu A/CAL/7/09, Day 182 | 161.9 [133.7 to 196.1] | 347.9 [254.0 to 476.5] | 154.0 [100.3 to 236.5] | 165.8 [131.9 to 208.5]

12. Secondary Outcome: Number of Seroconverted Subjects for HI Antibodies
Description: Seroconversion (SCR) was defined as follows:
  For initially seronegative subjects, antibody titer ≥ 1:40 after vaccination; For initially seropositive subjects, antibody titer after vaccination ≥ 4 fold the pre-vaccination antibody titer. The Flu strain assessed was Flu A/CAL/7/09, in subjects aged between 6 months to 9 years and 10 to 17 years, following the CHMP and the CBER guidance.
  The CHMP Criterion was fulfilled if the point estimate for SCR was > 40%. The CBER Criterion was fulfilled if the lower 97.5% confidence interval for SCR was > 40%.
Time Frame: At Day 21
Population: as for outcome 9
Measure: Number; unit: Subjects
Arm/Group | GSK2340274A_F1 6M-9Y Group | GSK2340274A_F2 10Y-17Y Group | GSK2340274A_F1 6M-35M Subgroup | GSK2340274A_F1 3Y-9Y Subgroup
Number analyzed (Participants) | 29 | 30 | 10 | 19
Subjects | 29 | 27 | 10 | 19

13. Secondary Outcome: Number of Seroconverted Subjects for HI Antibodies
Description: Seroconversion (SCR) was defined as follows:
  For initially seronegative subjects, antibody titer ≥ 1:40 after vaccination; For initially seropositive subjects, antibody titer after vaccination ≥ 4 fold the pre-vaccination antibody titer. The Flu strain assessed was Flu A/CAL/7/09, in subjects aged between 6 months to 9 years, following the CHMP and the CBER guidance.
  The CHMP Criterion was fulfilled if the point estimate for SCR was > 40%. The CBER Criterion was fulfilled if the lower 97.5% confidence interval for SCR was > 40%.
  Note: Analyses based on 95% CI for 10-17 year age category at Day 42 were not performed.
Time Frame: At Day 42
Population: as for outcome 10
Measure: Number; unit: Subjects
Arm/Group | GSK2340274A_F1 6M-35M Subgroup | GSK2340274A_F1 3Y-9Y Subgroup
Number analyzed (Participants) | 9 | 19
Subjects | 9 | 19

14. Secondary Outcome: Number of Seroconverted Subjects for HI Antibodies
Description: as for outcome 12
Time Frame: At Day 182
Population: as for outcome 8
Measure: Number; unit: Subjects
Arm/Group | GSK2340274A_F1 6M-9Y Group | GSK2340274A_F2 10Y-17Y Group | GSK2340274A_F1 6M-35M Subgroup | GSK2340274A_F1 3Y-9Y Subgroup
Number analyzed (Participants) | 28 | 29 | 9 | 19
Subjects | 27 | 26 | 9 | 18

15. Secondary Outcome: Number of Seroprotected Subjects for HI Antibodies
Description: A seroprotected subject was defined as a vaccinated subject with a serum hemagglutination inhibition (HI) titer equal to or above (≥) 1:40. The Flu strain assessed was Flu A/CAL/7/09, in subjects aged between 6 months to 9 years and 10 to 17 years, following the CHMP and the CBER guidance.
  The CHMP Criterion was fulfilled if the post-vaccination point estimate for SPR was > 70%.
  The CBER Criterion was fulfilled if the lower 97.5% confidence interval for SPR was > 70%.
Time Frame: At Days 0 and 21
Population: as for outcome 9
Measure: Number; unit: Subjects
Arm/Group | GSK2340274A_F1 6M-9Y Group | GSK2340274A_F2 10Y-17Y Group | GSK2340274A_F1 6M-35M Subgroup | GSK2340274A_F1 3Y-9Y Subgroup
Number analyzed (Participants) | 29 | 30 | 10 | 19
Subjects
  Flu A/CAL/7/09, Day 0 | 1 | 8 | 0 | 1
  Flu A/CAL/7/09, Day 21 | 29 | 29 | 10 | 19

16. Secondary Outcome: Number of Seroprotected Subjects for HI Antibodies
Description: A seroprotected subject was defined as a vaccinated subject with a serum HI titer equal to or above (≥) 1:40. The Flu strain assessed was Flu A/CAL/7/09, in subjects aged between 6 months to 9 years, following the CHMP and the CBER guidance.
  The CHMP Criterion was fulfilled if the post-vaccination point estimate for SPR was > 70%.
  The CBER Criterion was fulfilled if the lower 97.5% confidence interval for SPR was > 70%.
  Note: Analyses based on 95% CI for 10-17 year age category at Day 42 were not performed.
Time Frame: At Days 0 and 42
Population: as for outcome 10
Measure: Number; unit: Subjects
Arm/Group | GSK2340274A_F1 6M-35M Subgroup | GSK2340274A_F1 3Y-9Y Subgroup
Number analyzed (Participants) | 9 | 19
Subjects
  Flu A/CAL/7/09, Day 0 | 0 | 1
  Flu A/CAL/7/09, Day 42 | 9 | 19

17. Secondary Outcome: Number of Seroprotected Subjects for HI Antibodies
Description: A seroprotected subject was defined as a vaccinated subject with a serum HI titer equal to or above (≥) 1:40. The Flu strain assessed was Flu A/CAL/7/09, in subjects aged between 6 months to 9 years and 10 to 17 years, following the CHMP and the CBER guidance.
  The CHMP Criterion was fulfilled if the post-vaccination point estimate for SPR was > 70%.
  The CBER Criterion was fulfilled if the lower 97.5% confidence interval for SPR was > 70%.
Time Frame: At Days 0 and 182
Population: as for outcome 8
Measure: Number; unit: Subjects
Arm/Group | GSK2340274A_F1 6M-9Y Group | GSK2340274A_F2 10Y-17Y Group | GSK2340274A_F1 6M-35M Subgroup | GSK2340274A_F1 3Y-9Y Subgroup
Number analyzed (Participants) | 28 | 29 | 9 | 19
Subjects
  Flu A/CAL/7/09, Day 0 | 1 | 7 | 0 | 1
  Flu A/CAL/7/09, Day 182 | 28 | 29 | 9 | 19

18. Secondary Outcome: Seroconversion Factor (SCF) for HI Antibodies Against Flu A/CAL/7/09 Strain of Influenza Disease
Description: Seroconversion factor (SCF) was defined as the fold increase in serum HI GMTs post-vaccination compared to pre-vaccination. The Flu strain assessed was Flu A/CAL/7/09, in subjects aged between 6 months to 9 years and 10 to 17 years, following the CHMP guidance.
  The CHMP Criterion was fulfilled if the point estimate for SCF was > 2.5.
Time Frame: At Day 21
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | GSK2340274A_F1 6M-9Y Group | GSK2340274A_F2 10Y-17Y Group | GSK2340274A_F1 6M-35M Subgroup | GSK2340274A_F1 3Y-9Y Subgroup
Number analyzed (Participants) | 29 | 30 | 10 | 19
Titers | 27.1 [20.4 to 36.1] | 22.1 [13.6 to 35.9] | 23.5 [14.4 to 38.2] | 29.3 [19.9 to 42.9]

19. Secondary Outcome: SCF for HI Antibodies Against Flu A/CAL/7/09 Strain of Influenza Disease
Description: SCF was defined as the fold increase in serum HI GMTs post-vaccination compared to pre-vaccination. The Flu strain assessed was Flu A/CAL/7/09, in subjects aged between 6 months to 9 years, following the CHMP guidance.
  The CHMP Criterion was fulfilled if the point estimate for SCF was > 2.5. Note: Analyses based on 95% CI for 10-17 year age category at Day 42 were not performed.
Time Frame: At Day 42
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | GSK2340274A_F1 6M-35M Subgroup | GSK2340274A_F1 3Y-9Y Subgroup
Number analyzed (Participants) | 9 | 19
Titers | 256.0 [161.4 to 406.1] | 112.8 [74.6 to 170.5]

20. Secondary Outcome: SCF for HI Antibodies Against Flu A/CAL/7/09 Strain of Influenza Disease
Description: SCF was defined as the fold increase in serum HI GMTs post-vaccination compared to pre-vaccination. The Flu strain assessed was Flu A/CAL/7/09, in subjects aged between 6 months to 9 years and 10 to 17 years, following the CHMP guidance.
  The CHMP Criterion was fulfilled if the point estimate for SCF was > 2.5.
Time Frame: At Day 182
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | GSK2340274A_F1 6M-9Y Group | GSK2340274A_F2 10Y-17Y Group | GSK2340274A_F1 6M-35M Subgroup | GSK2340274A_F1 3Y-9Y Subgroup
Number analyzed (Participants) | 28 | 29 | 9 | 19
Titers | 25.3 [18.4 to 34.7] | 23.5 [14.9 to 37.1] | 30.8 [20.1 to 47.3] | 23.1 [14.9 to 35.8]

21. Secondary Outcome: Number of Subjects With Neutralizing Antibody Concentrations Above the Cut-off Value
Description: The cut-off values for the humoral immune response in terms of vaccine neutralizing antibodies were equal to or above (≥) 1:8. The Flu strain assessed was Flu A/Neth/602/09 H1N1, in subjects aged between 6 months to 9 years and 10 to 17 years, following the CHMP and the CBER guidance.
Time Frame: At Days 0 and 21
Population: The analysis was performed on the ATP cohort for immunogenicity at Day 21, which included all evaluable subjects for whom assay results for antibodies against Flu A/Neth/602/09 H1N1 antigen for the blood sample taken 21 days after the first vaccination were available.
Measure: Number; unit: Subjects
Arm/Group | GSK2340274A_F1 6M-9Y Group | GSK2340274A_F2 10Y-17Y Group
Number analyzed (Participants) | 29 | 30
Subjects
  Flu A/Neth/602/09 H1N1, Day 0 (N=29;30) | 3 | 14
  Flu A/Neth/602/09 H1N1, Day 21 (N=29;29) | 28 | 28

22. Secondary Outcome: Number of Subjects With Neutralizing Antibody Concentrations Above the Cut-off Value
Description: as for outcome 21
Time Frame: At Days 0 and 42
Population: The analysis was performed on the ATP cohort for immunogenicity at Day 42, which included all evaluable subjects for whom assay results for antibodies against Flu A/Neth/602/09 H1N1 antigen for the blood samples taken on Day 42 (21 days after the second vaccination) were available.
Measure: Number; unit: Subjects
Arm/Group | GSK2340274A_F1 6M-9Y Group | GSK2340274A_F2 10Y-17Y Group
Number analyzed (Participants) | 28 | 30
Subjects
  Flu A/Neth/602/09 H1N1, Day 0 | 3 | 14
  Flu A/Neth/602/09 H1N1, Day 42 | 28 | 30

23. Secondary Outcome: Number of Subjects With Neutralizing Antibody Concentrations Above the Cut-off Value
Description: as for outcome 21
Time Frame: At Days 0 and 182
Population: The analysis was performed on the ATP cohort for immunogenicity at Day 182, which included all evaluable subjects for whom assay results for antibodies against Flu A/Neth/602/09 H1N1 antigen for the blood samples taken on Day 182 were available.
Measure: Number; unit: Subjects
Arm/Group | GSK2340274A_F1 6M-9Y Group | GSK2340274A_F2 10Y-17Y Group
Number analyzed (Participants) | 28 | 29
Subjects
  Flu A/Neth/602/09 H1N1, Day 0 | 3 | 13
  Flu A/Neth/602/09 H1N1, Day 182 | 28 | 29

24. Secondary Outcome: Titers for Serum Neutralizing Antibodies Against Flu A/Neth/602/09 Strain of Influenza Disease
Description: Titers are presented as geometric mean titers (GMTs). The reference seropositivity cut-off value was ≥ 1:8. The Flu strain assessed was Flu A/Neth/602/09 H1N1, in subjects aged between 6 months to 9 years and 10 to 17 years, following the CHMP and the CBER guidance.
Time Frame: At Days 0 and 21
Population: as for outcome 21
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | GSK2340274A_F1 6M-9Y Group | GSK2340274A_F2 10Y-17Y Group
Number analyzed (Participants) | 29 | 30
Titers
  Flu A/Neth/602/09 H1N1, Day 0 (N=29;30) | 4.9 [3.7 to 6.5] | 11.3 [6.8 to 18.9]
  Flu A/Neth/602/09 H1N1, Day 21 (N=29;29) | 53.8 [31.2 to 92.7] | 121.2 [68.4 to 214.9]

25. Secondary Outcome: Titers for Serum Neutralizing Antibodies Against Flu A/Neth/602/09 Strain of Influenza Disease
Description: as for outcome 24
Time Frame: At Days 0 and 42
Population: as for outcome 22
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | GSK2340274A_F1 6M-9Y Group | GSK2340274A_F2 10Y-17Y Group
Number analyzed (Participants) | 28 | 30
Titers
  Flu A/Neth/602/09 H1N1, Day 0 | 4.9 [3.7 to 6.6] | 11.3 [6.8 to 18.9]
  Flu A/Neth/602/09 H1N1, Day 42 | 551.1 [417.0 to 728.5] | 702.4 [433.5 to 1138.0]

26. Secondary Outcome: Titers for Serum Neutralizing Antibodies Against Flu A/Neth/602/09 Strain of Influenza Disease
Description: as for outcome 24
Time Frame: At Days 0 and 182
Population: as for outcome 23
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | GSK2340274A_F1 6M-9Y Group | GSK2340274A_F2 10Y-17Y Group
Number analyzed (Participants) | 28 | 29
Titers
  Flu A/Neth/602/09 H1N1, Day 0 | 4.9 [3.7 to 6.6] | 11.4 [6.7 to 19.4]
  Flu A/Neth/602/09 H1N1, Day 182 | 149.6 [104.7 to 213.6] | 213.3 [141.7 to 321.0]

27. Secondary Outcome: Number of Subjects With Vaccine Response Rates (VRR) for Neutralizing Antibodies Against Flu A/Neth/602/09 H1N1
Description: VRR is defined as the number of vaccinees that have a 4-fold increase between pre- and post-vaccination titers. The Flu strain assessed was Flu A/Neth/602/09 H1N1, in subjects aged between 6 months to 9 years and 10 to 17 years, following the CHMP and the CBER guidance.
Time Frame: At Day 21
Population: as for outcome 21
Measure: Number; unit: Subjects
Arm/Group | GSK2340274A_F1 6M-9Y Group | GSK2340274A_F2 10Y-17Y Group
Number analyzed (Participants) | 29 | 29
Subjects | 15 | 17

28. Secondary Outcome: Number of Subjects With Vaccine Response Rates (VRR) for Neutralising Antibodies Against Flu A/Neth/602/09 H1N1
Description: as for outcome 27
Time Frame: At Day 42
Population: as for outcome 22
Measure: Number; unit: Subjects
Arm/Group | GSK2340274A_F1 6M-9Y Group | GSK2340274A_F2 10Y-17Y Group
Number analyzed (Participants) | 28 | 30
Subjects | 28 | 30

29. Secondary Outcome: Number of Subjects With Vaccine Response Rates (VRR) for Neutralising Antibodies Against Flu A/Neth/602/09 H1N1
Description: as for outcome 27
Time Frame: At Day 182
Population: as for outcome 23
Measure: Number; unit: Subjects
Arm/Group | GSK2340274A_F1 6M-9Y Group | GSK2340274A_F2 10Y-17Y Group
Number analyzed (Participants) | 28 | 29
Subjects | 27 | 24

30. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain [child below (<) 6 years] = cried when limb was moved/spontaneously painful. Grade 3 pain [child equal to or above (≥) 6 years] = pain that prevented normal activity. Grade 3 redness/swelling = redness/swelling spreading beyond 100 millimeters (mm) of injection site.
Time Frame: During the 7-day (Days 0-6) post-vaccination period following each dose and across doses
Population: The analysis was performed on The Total Vaccinated Cohort which included all vaccinated subjects.
Measure: Number; unit: Subjects
Groups:
- GSK2340274A_F1 6M-5Y Subgroup: Healthy male or female Japanese children, between and including 6 months to 5 years of age, who received two doses of GSK2340274A vaccine (formulation 1), administered intramuscularly into the deltoid region of the arm (intramuscularly into the anterolateral part of the thigh for subjects below 12 months of age at the entry of the study), according to 0, 21-day schedule.
- GSK2340274A_F1 6Y-9Y Subgroup: Healthy male or female Japanese children, between and including 6 to 9 years of age, who received two doses of GSK2340274A vaccine (formulation 1), administered intramuscularly into the deltoid region of the arm, according to 0, 21-day schedule.
Arm/Group | GSK2340274A_F1 6M-5Y Subgroup | GSK2340274A_F1 6Y-9Y Subgroup | GSK2340274A_F2 10Y-17Y Group
Number analyzed (Participants) | 24 | 6 | 30
Subjects
  Any Pain, Dose 1 (N=24;6;30) | 19 | 5 | 30
  Grade 3 Pain, Dose 1 (N=24;6;30) | 1 | 0 | 3
  Any Redness, Dose 1 (N=24;6;30) | 0 | 1 | 7
  Grade 3 Redness, Dose 1 (N=24;6;30) | 0 | 0 | 0
  Any Swelling, Dose 1 (N=24;6;30) | 5 | 2 | 14
  Grade 3 Swelling, Dose 1 (N=24;6;30) | 0 | 0 | 1
  Any Pain, Dose 2 (N=23;6;30) | 16 | 5 | 30
  Grade 3 Pain, Dose 2 (N=23;6;30) | 1 | 0 | 2
  Any Redness, Dose 2 (N=23;6;30) | 2 | 0 | 5
  Grade 3 Redness, Dose 2 (N=23;6;30) | 0 | 0 | 0
  Any Swelling, Dose 2 (N=23;6;30) | 4 | 2 | 15
  Grade 3 Swelling, Dose 2 (N=23;6;30) | 0 | 0 | 1
  Any Pain, Across Doses (N=24;6;30) | 19 | 6 | 30
  Grade 3 Pain, Across Doses (N=24;6;30) | 2 | 0 | 5
  Any Redness, Across Doses (N=24;6;30) | 2 | 1 | 10
  Grade 3 Redness, Across Doses (N=24;6;30) | 0 | 0 | 0
  Any Swelling, Across Doses (N=24;6;30) | 8 | 2 | 16
  Grade 3 Swelling, Across Doses (N=24;6;30) | 0 | 0 | 2

31. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Assessed solicited general symptoms were drowsiness, irritability, loss of appetite, fever [defined as axillary temperature equal to or above (≥) 37.5 degrees Celsius (°C)]. Any = occurrence of any general symptoms regardless of their intensity grade or their relation to vaccination. Grade 3 symptom = symptom that prevented normal activity. Grade 3 loss of appetite = not eating at all. Grade 3 fever = fever ≥ 39.0 °C - ≤ 40.0°C. Related = symptom assessed by the investigator as causally related to the vaccination.
Time Frame: During the 7-day (Days 0-6) post-vaccination period following each dose and across doses
Population: The analysis was performed on the Total Vaccinated Cohort which included all vaccinated subjects.
Measure: Number; unit: Subjects
Arm/Group | GSK2340274A_F1 6M-5Y Subgroup
Number analyzed (Participants) | 24
Subjects
  Any Drowsiness, Dose 1 (N=24) | 5
  Grade 3 Drowsiness, Dose 1 (N=24) | 0
  Related Drowsiness, Dose 1 (N=24) | 5
  Any Irritability, Dose 1 (N=24) | 6
  Grade 3 Irritability, Dose 1 (N=24) | 1
  Related Irritability, Dose 1 (N=24) | 6
  Any Loss of appetite, Dose 1 (N=24) | 5
  Grade 3 Loss of appetite, Dose 1 (N=24) | 0
  Related Loss of appetite, Dose 1 (N=24) | 4
  Any Fever, Dose 1 (N=24) | 3
  Grade 3 Fever, Dose 1 (N=24) | 0
  Related Fever, Dose 1 (N=24) | 3
  Any Drowsiness, Dose 2 (N=23) | 7
  Grade 3 Drowsiness, Dose 2 (N=23) | 0
  Related Drowsiness, Dose 2 (N=23) | 7
  Any Irritability, Dose 2 (N=23) | 6
  Grade 3 Irritability, Dose 2 (N=23) | 0
  Related Irritability, Dose 2 (N=23) | 5
  Any Loss of appetite, Dose 2 (N=23) | 5
  Grade 3 Loss of appetite, Dose 2 (N=23) | 1
  Related Loss of appetite, Dose 2 (N=23) | 5
  Any Fever, Dose 2 (N=23) | 6
  Grade 3 Fever, Dose 2 (N=23) | 2
  Related Fever, Dose 2 (N=23) | 5
  Any Drowsiness, Across doses (N=24) | 8
  Grade 3 Drowsiness, Across doses (N=24) | 0
  Related Drowsiness, Across doses (N=24) | 8
  Any Irritability, Across doses (N=24) | 8
  Grade 3 Irritability, Across doses (N=24) | 1
  Related Irritability, Across doses (N=24) | 7
  Any Loss of appetite, Across doses (N=24) | 7
  Grade 3 Loss of appetite, Across doses (N=24) | 1
  Related Loss of appetite, Across doses (N=24) | 6
  Any Fever, Across doses (N=24) | 8
  Grade 3 Fever, Across doses (N=24) | 2
  Related Fever, Across doses (N=24) | 7

32. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Assessed solicited general symptoms were fatigue, gastrointestinal, headache, joint pain at other location, muscle aches, shivering, sweating, and fever [defined as axillary temperature equal to or above 37.5 degrees Celsius (°C)]. Any = occurrence of any general symptoms regardless of their intensity grade or their relation to vaccination. Grade 3 symptom = symptom that prevented normal activity. Grade 3 fever = fever ≥ 39.0°C - ≤ 40.0°C. Related symptom = symptom assessed by the investigator as causally related to the study vaccination.
Time Frame: During the 7-day (Days 0-6) post-vaccination period following each dose and across doses
Population: The analysis was performed on the Total Vaccinated Cohort which included all vaccinated subjects.
Measure: Number; unit: Subjects
Arm/Group | GSK2340274A_F1 6Y-9Y Subgroup | GSK2340274A_F2 10Y-17Y Group
Number analyzed (Participants) | 6 | 30
Subjects
  Any Fatigue, Dose 1 | 1 | 11
  Grade 3 Fatigue, Dose 1 | 0 | 1
  Related Fatigue, Dose 1 | 0 | 10
  Any Gastrointestinal, Dose 1 | 1 | 3
  Grade 3 Gastrointestinal, Dose 1 | 0 | 0
  Related Gastrointestinal, Dose 1 | 0 | 3
  Any Headache, Dose 1 | 2 | 12
  Grade 3 Headache, Dose 1 | 0 | 0
  Related Headache, Dose 1 | 0 | 11
  Any Joint pain, Dose 1 | 0 | 5
  Grade 3 Joint pain, Dose 1 | 0 | 0
  Related Joint pain, Dose 1 | 0 | 4
  Any Muscle aches, Dose 1 | 0 | 7
  Grade 3 Muscle aches, Dose 1 | 0 | 0
  Related Muscle aches, Dose 1 | 0 | 7
  Any Shivering, Dose 1 | 1 | 7
  Grade 3 Shivering, Dose 1 | 0 | 0
  Related Shivering, Dose 1 | 1 | 6
  Any Sweating, Dose 1 | 0 | 2
  Grade 3 Sweating, Dose 1 | 0 | 1
  Related Sweating, Dose 1 | 0 | 1
  Any Fever, Dose 1 | 2 | 4
  Grade 3 Fever, Dose 1 | 0 | 3
  Related Fever, Dose 1 | 1 | 3
  Any Fatigue, Dose 2 | 1 | 11
  Grade 3 Fatigue, Dose 2 | 0 | 1
  Related Fatigue, Dose 2 | 1 | 11
  Any Gastrointestinal, Dose 2 | 1 | 3
  Grade 3 Gastrointestinal, Dose 2 | 0 | 0
  Related Gastrointestinal, Dose 2 | 1 | 3
  Any Headache, Dose 2 | 1 | 17
  Grade 3 Headache, Dose 2 | 0 | 2
  Related Headache, Dose 2 | 1 | 16
  Any Joint pain, Dose 2 | 0 | 7
  Grade 3 Joint pain, Dose 2 | 0 | 0
  Related Joint pain, Dose 2 | 0 | 6
  Any Muscle aches, Dose 2 | 0 | 9
  Grade 3 Muscle aches, Dose 2 | 0 | 0
  Related Muscle aches, Dose 2 | 0 | 8
  Any Shivering, Dose 2 | 0 | 8
  Grade 3 Shivering, Dose 2 | 0 | 0
  Related Shivering, Dose 2 | 0 | 8
  Any Sweating, Dose 2 | 0 | 3
  Grade 3 Sweating, Dose 2 | 0 | 0
  Related Sweating, Dose 2 | 0 | 3
  Any Fever, Dose 2 | 0 | 7
  Grade 3 Fever, Dose 2 | 0 | 0
  Related Fever, Dose 2 | 0 | 7
  Any Fatigue, Across doses | 2 | 14
  Grade 3 Fatigue, Across doses | 0 | 2
  Related Fatigue, Across doses | 1 | 14
  Any Gastrointestinal, Across doses | 2 | 4
  Grade 3 Gastrointestinal, Across doses | 0 | 0
  Related Gastrointestinal, Across doses | 1 | 4
  Any Headache, Across doses | 3 | 20
  Grade 3 Headache, Across doses | 0 | 2
  Related Headache, Across doses | 1 | 19
  Any Joint pain, Across doses | 0 | 9
  Grade 3 Joint pain, Across doses | 0 | 0
  Related Joint pain, Across doses | 0 | 8
  Any Muscle aches, Across doses | 0 | 11
  Grade 3 Muscle aches, Across doses | 0 | 0
  Related Muscle aches, Across doses | 0 | 10
  Any Shivering, Across doses | 1 | 11
  Grade 3 Shivering, Across doses | 0 | 0
  Related Shivering, Across doses | 1 | 11
  Any Sweating, Across doses | 0 | 5
  Grade 3 Sweating, Across doses | 0 | 1
  Related Sweating, Across doses | 0 | 4
  Any Fever, Across doses | 2 | 8
  Grade 3 Fever, Across doses | 0 | 3
  Related Fever, Across doses | 1 | 8

33. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination. Grade 3 AE = an AE which prevented normal, everyday activities. Related = AE assessed by the investigator as related to the vaccination.
Time Frame: Up to 84 days (Days 0-83) after the first vaccination
Population: The analysis was performed on the Total Vaccinated Cohort which included all vaccinated subjects.
Measure: Number; unit: Subjects
Arm/Group | GSK2340274A_F1 6M-9Y Group | GSK2340274A_F2 10Y-17Y Group
Number analyzed (Participants) | 30 | 30
Subjects
  Any AE(s) | 19 | 21
  Grade 3 AE(s) | 9 | 7
  Related AE(s) | 9 | 8

34. Secondary Outcome: Number of Subjects With Medically Attended Events (MAEs)
Description: MAEs were defined as events for which the subject received medical attention defined as hospitalization, an emergency room visit, or a visit to or from medical personnel (medical doctor) for any reason. Any MAE(s) = occurrence of any MAE(s) regardless of intensity grade or relation to vaccination. Analysis of intensity and relationship to vaccination of MAEs was not performed.
Time Frame: During the entire study period (from Day 0 to Day 182)
Population: The analysis was performed on the Total Vaccinated Cohort which included all vaccinated subjects.
Measure: Number; unit: Subjects
Arm/Group | GSK2340274A_F1 6M-5Y Subgroup | GSK2340274A_F1 6Y-9Y Subgroup | GSK2340274A_F2 10Y-17Y Group
Number analyzed (Participants) | 24 | 6 | 30
Subjects | 14 | 2 | 10

35. Secondary Outcome: Number of Subjects With Potential Immune-Mediated Diseases (pIMDs)
Description: Potential immune-mediated diseases (pIMDs) are a subset of AEs that include autoimmune diseases and other inflammatory and/or neurologic disorders of interest which may or may not have an autoimmune aetiology.
Time Frame: During the entire study period (from Day 0 to Day 182)
Population: The analysis was performed on the Total Vaccinated Cohort which included all vaccinated subjects.
Measure: Number; unit: Subjects
Arm/Group | GSK2340274A_F1 6M-5Y Subgroup | GSK2340274A_F1 6Y-9Y Subgroup | GSK2340274A_F2 10Y-17Y Group
Number analyzed (Participants) | 24 | 6 | 30
Subjects | 0 | 0 | 0

36. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life-threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: During the entire study period (from Day 0 to Day 182)
Population: The analysis was performed on the Total Vaccinated Cohort which included all vaccinated subjects.
Measure: Number; unit: Subjects
Arm/Group | GSK2340274A_F1 6M-9Y Group | GSK2340274A_F2 10Y-17Y Group
Number analyzed (Participants) | 30 | 30
Subjects | 1 | 1

37. Secondary Outcome: Number of Subjects With Normal or Abnormal Biochemical Levels
Description: Among biochemical parameters assessed were Alanine Amino Transferase (ALAT), Albumin, Alkaline Phosphatase (AP), Aspartate Amino Transferase (ASAT), Bilirubin, Bilirubin Conjugated/Direct, Cholesterol, Chloride, Creatinine, Creatine Phosphokinase (CK), Gamma-Glutamyl Transpeptidase (GGT), Potassium, Lactate dehydrogenase (LDH), Sodium, Protein, Urate/Uric acid and Blood Urea Nitrogen (BUN).
  Unknown = value unknown for the specified time point and laboratory parameter; Below = value below the laboratory reference range defined for the specified time point and laboratory parameter; Within = value within the laboratory reference range defined for the specified time point and laboratory parameter; Above = value above the laboratory reference range defined for the specified time point and laboratory parameter.
Time Frame: At Days 0, 7 and 42
Population: The analysis was performed on the Total Vaccinated Cohort which included all vaccinated subjects.
Measure: Number; unit: Subjects
Arm/Group | GSK2340274A_F1 6M-5Y Subgroup | GSK2340274A_F1 6Y-9Y Subgroup | GSK2340274A_F2 10Y-17Y Group
Number analyzed (Participants) | 23 | 6 | 30
Subjects
  ALAT Unknown, Day 0 (N=22;6;29) | 0 | 0 | 0
  ALAT Unknown, Day 7 (N=23;6;30) | 0 | 0 | 0
  ALAT Unknown, Day 42 (N=22;6;30) | 0 | 0 | 0
  ALAT Below, Day 0 (N=22;6;29) | 0 | 0 | 0
  ALAT Below, Day 7 (N=23;6;30) | 0 | 0 | 0
  ALAT Below, Day 42 (N=22;6;30) | 0 | 0 | 0
  ALAT Within, Day 0 (N=22;6;29) | 22 | 6 | 28
  ALAT Within, Day 7 (N=23;6;30) | 23 | 6 | 28
  ALAT Within, Day 42 (N=22;6;30) | 22 | 6 | 30
  ALAT Above, Day 0 (N=22;6;29) | 0 | 0 | 1
  ALAT Above, Day 7 (N=23;6;30) | 0 | 0 | 2
  ALAT Above, Day 42 (N=22;6;30) | 0 | 0 | 0
  Albumin Unknown, Day 0 (N=22;6;29) | 0 | 0 | 0
  Albumin Unknown, Day 7 (N=23;6;30) | 0 | 0 | 0
  Albumin Unknown, Day 42 (N=22;6;30) | 0 | 0 | 0
  Albumin Below, Day 0 (N=22;6;29) | 0 | 0 | 0
  Albumin Below, Day 7 (N=23;6;30) | 0 | 0 | 0
  Albumin Below, Day 42 (N=22;6;30) | 2 | 0 | 1
  Albumin Within, Day 0 (N=22;6;29) | 21 | 6 | 27
  Albumin Within, Day 7 (N=23;6;30) | 22 | 6 | 29
  Albumin Within, Day 42 (N=22;6;30) | 19 | 6 | 28
  Albumin Above, Day 0 (N=22;6;29) | 1 | 0 | 2
  Albumin Above, Day 7 (N=23;6;30) | 1 | 0 | 1
  Albumin Above, Day 42 (N=22;6;30) | 1 | 0 | 1
  AP Unknown, Day 0 (N=22;6;29) | 0 | 0 | 0
  AP Unknown, Day 7 (N=23;6;30) | 0 | 0 | 0
  AP Unknown, Day 42 (N=22;6;30) | 1 | 0 | 0
  AP Below, Day 0 (N=22;6;29) | 0 | 0 | 0
  AP Below, Day 7 (N=23;6;30) | 0 | 0 | 0
  AP Below, Day 42 (N=22;6;30) | 0 | 0 | 0
  AP Within, Day 0 (N=22;6;29) | 0 | 0 | 8
  AP Within, Day 7 (N=23;6;30) | 0 | 0 | 9
  AP Within, Day 42 (N=22;6;30) | 0 | 0 | 9
  AP Above, Day 0 (N=22;6;29) | 22 | 6 | 21
  AP Above, Day 7 (N=23;6;30) | 23 | 6 | 21
  AP Above, Day 42 (N=22;6;30) | 21 | 6 | 21
  ASAT Unknown, Day 0 (N=22;6;29) | 0 | 0 | 0
  ASAT Unknown, Day 7 (N=23;6;30) | 0 | 0 | 0
  ASAT Unknown, Day 42 (N=22;6;30) | 1 | 0 | 0
  ASAT Below, Day 0 (N=22;6;29) | 0 | 0 | 1
  ASAT Below, Day 7 (N=23;6;30) | 0 | 0 | 0
  ASAT Below, Day 42 (N=22;6;30) | 0 | 0 | 0
  ASAT Within, Day 0 (N=22;6;29) | 21 | 6 | 27
  ASAT Within, Day 7 (N=23;6;30) | 21 | 6 | 30
  ASAT Within, Day 42 (N=22;6;30) | 20 | 6 | 30
  ASAT Above, Day 0 (N=22;6;29) | 1 | 0 | 1
  ASAT Above, Day 7 (N=23;6;30) | 2 | 0 | 0
  ASAT Above, Day 42 (N=22;6;30) | 1 | 0 | 0
  Bilirubin Unknown, Day 0 (N=22;6;29) | 0 | 0 | 0
  Bilirubin Unknown, Day 7 (N=23;6;30) | 0 | 0 | 0
  Bilirubin Unknown, Day 42 (N=22;6;30) | 0 | 0 | 0
  Bilirubin Below, Day 0 (N=22;6;29) | 0 | 0 | 0
  Bilirubin Below, Day 7 (N=23;6;30) | 0 | 0 | 0
  Bilirubin Below, Day 42 (N=22;6;30) | 0 | 0 | 0
  Bilirubin Within, Day 0 (N=22;6;29) | 22 | 6 | 29
  Bilirubin Within, Day 7 (N=23;6;30) | 23 | 6 | 30
  Bilirubin Within, Day 42 (N=22;6;30) | 22 | 6 | 29
  Bilirubin Above, Day 0 (N=22;6;29) | 0 | 0 | 0
  Bilirubin Above, Day 7 (N=23;6;30) | 0 | 0 | 0
  Bilirubin Above, Day 42 (N=22;6;30) | 0 | 0 | 1
  Bilirubin Conj./Direct Unknown, Day 0 (N=22;6;29) | 0 | 0 | 0
  Bilirubin Conj./Direct Unknown, Day 7 (N=23;6;30) | 0 | 0 | 0
  Bilirubin Conj./Direct Unknown, Day 42 (N=22;6;30) | 0 | 0 | 0
  Bilirubin Conj./Direct Below, Day 0 (N=22;6;29) | 0 | 0 | 0
  Bilirubin Conj./Direct Below, Day 7 (N=23;6;30) | 0 | 0 | 0
  Bilirubin Conj./Direct Below, Day 42 (N=22;6;30) | 0 | 0 | 0
  Bilirubin Conj./Direct Within, Day 0 (N=22;6;29) | 22 | 6 | 28
  Bilirubin Conj./Direct Within, Day 7 (N=23;6;30) | 23 | 6 | 30
  Bilirubin Conj./Direct Within, Day 42 (N=22;6;30) | 22 | 6 | 27
  Bilirubin Conj./Direct Above, Day 0 (N=22;6;29) | 0 | 0 | 1
  Bilirubin Conj./Direct Above, Day 7 (N=23;6;30) | 0 | 0 | 0
  Bilirubin Conj./Direct Above, Day 42 (N=22;6;30) | 0 | 0 | 3
  Cholesterol Unknown, Day 0 (N=22;6;29) | 0 | 0 | 0
  Cholesterol Unknown, Day 7 (N=23;6;30) | 0 | 0 | 0
  Cholesterol Unknown, Day 42 (N=22;6;30) | 0 | 0 | 0
  Cholesterol Below, Day 0 (N=22;6;29) | 7 | 2 | 9
  Cholesterol Below, Day 7 (N=23;6;30) | 8 | 2 | 12
  Cholesterol Below, Day 42 (N=22;6;30) | 8 | 2 | 10
  Cholesterol Within, Day 0 (N=22;6;29) | 13 | 4 | 20
  Cholesterol Within, Day 7 (N=23;6;30) | 14 | 4 | 18
  Cholesterol Within, Day 42 (N=22;6;30) | 14 | 4 | 19
  Cholesterol Above, Day 0 (N=22;6;29) | 2 | 0 | 0
  Cholesterol Above, Day 7 (N=23;6;30) | 1 | 0 | 0
  Cholesterol Above, Day 42 (N=22;6;30) | 0 | 0 | 1
  Chloride Unknown, Day 0 (N=22;6;29) | 0 | 0 | 0
  Chloride Unknown, Day 7 (N=23;6;30) | 0 | 0 | 0
  Chloride Unknown, Day 42 (N=22;6;30) | 0 | 0 | 0
  Chloride Below, Day 0 (N=22;6;29) | 0 | 0 | 0
  Chloride Below, Day 7 (N=23;6;30) | 0 | 0 | 0
  Chloride Below, Day 42 (N=22;6;30) | 0 | 0 | 0
  Chloride Within, Day 0 (N=22;6;29) | 22 | 6 | 29
  Chloride Within, Day 7 (N=23;6;30) | 23 | 6 | 29
  Chloride Within, Day 42 (N=22;6;30) | 22 | 6 | 29
  Chloride Above, Day 0 (N=22;6;29) | 0 | 0 | 0
  Chloride Above, Day 7 (N=23;6;30) | 0 | 0 | 1
  Chloride Above, Day 42 (N=22;6;30) | 0 | 0 | 1
  Creatinine Unknown, Day 0 (N=22;6;29) | 0 | 0 | 0
  Creatinine Unknown, Day 7 (N=23;6;30) | 0 | 0 | 0
  Creatinine Unknown, Day 42 (N=22;6;30) | 0 | 0 | 0
  Creatinine Below, Day 0 (N=22;6;29) | 22 | 6 | 11
  Creatinine Below, Day 7 (N=23;6;30) | 23 | 6 | 8
  Creatinine Below, Day 42 (N=22;6;30) | 22 | 6 | 12
  Creatinine Within, Day 0 (N=22;6;29) | 0 | 0 | 18
  Creatinine Within, Day 7 (N=23;6;30) | 0 | 0 | 22
  Creatinine Within, Day 42 (N=22;6;30) | 0 | 0 | 18
  Creatinine Above, Day 0 (N=22;6;29) | 0 | 0 | 0
  Creatinine Above, Day 7 (N=23;6;30) | 0 | 0 | 0
  Creatinine Above, Day 42 (N=22;6;30) | 0 | 0 | 0
  CK Unknown, Day 0 (N=22;6;29) | 0 | 0 | 0
  CK Unknown, Day 7 (N=23;6;30) | 0 | 0 | 0
  CK Unknown, Day 42 (N=22;6;30) | 0 | 0 | 0
  CK Below, Day 0 (N=22;6;29) | 0 | 0 | 0
  CK Below, Day 7 (N=23;6;30) | 0 | 0 | 0
  CK Below, Day 42 (N=22;6;30) | 0 | 0 | 0
  CK Within, Day 0 (N=22;6;29) | 17 | 6 | 28
  CK Within, Day 7 (N=23;6;30) | 19 | 6 | 28
  CK Within, Day 42 (N=22;6;30) | 20 | 5 | 27
  CK Above, Day 0 (N=22;6;29) | 5 | 0 | 1
  CK Above, Day 7 (N=23;6;30) | 4 | 0 | 2
  CK Above, Day 42 (N=22;6;30) | 2 | 1 | 3
  GGT Unknown, Day 0 (N=22;6;29) | 0 | 0 | 0
  GGT Unknown, Day 7 (N=23;6;30) | 0 | 0 | 0
  GGT Unknown, Day 42 (N=22;6;30) | 0 | 0 | 0
  GGT Below, Day 0 (N=22;6;29) | 0 | 0 | 0
  GGT Below, Day 7 (N=23;6;30) | 0 | 0 | 0
  GGT Below, Day 42 (N=22;6;30) | 0 | 0 | 0
  GGT Within, Day 0 (N=22;6;29) | 22 | 6 | 29
  GGT Within, Day 7 (N=23;6;30) | 23 | 6 | 29
  GGT Within, Day 42 (N=22;6;30) | 22 | 6 | 29
  GGT Above, Day 0 (N=22;6;29) | 0 | 0 | 0
  GGT Above, Day 7 (N=23;6;30) | 0 | 0 | 1
  GGT Above, Day 42 (N=22;6;30) | 0 | 0 | 1
  Potassium Unknown, Day 0 (N=22;6;29) | 0 | 0 | 0
  Potassium Unknown, Day 7 (N=23;6;30) | 0 | 0 | 0
  Potassium Unknown, Day 42 (N=22;6;30) | 1 | 0 | 0
  Potassium Below, Day 0 (N=22;6;29) | 0 | 0 | 0
  Potassium Below, Day 7 (N=23;6;30) | 0 | 0 | 0
  Potassium Below, Day 42 (N=22;6;30) | 0 | 0 | 0
  Potassium Within, Day 0 (N=22;6;29) | 21 | 6 | 29
  Potassium Within, Day 7 (N=23;6;30) | 23 | 6 | 30
  Potassium Within, Day 42 (N=22;6;30) | 20 | 6 | 30
  Potassium Above, Day 0 (N=22;6;29) | 1 | 0 | 0
  Potassium Above, Day 7 (N=23;6;30) | 0 | 0 | 0
  Potassium Above, Day 42 (N=22;6;30) | 1 | 0 | 0
  LDH Unknown, Day 0 (N=22;6;29) | 0 | 0 | 0
  LDH Unknown, Day 7 (N=23;6;30) | 0 | 0 | 0
  LDH Unknown, Day 42 (N=22;6;30) | 1 | 0 | 0
  LDH Below, Day 0 (N=22;6;29) | 0 | 0 | 0
  LDH Below, Day 7 (N=23;6;30) | 0 | 0 | 0
  LDH Below, Day 42 (N=22;6;30) | 0 | 0 | 0
  LDH Within, Day 0 (N=22;6;29) | 4 | 2 | 26
  LDH Within, Day 7 (N=23;6;30) | 2 | 2 | 29
  LDH Within, Day 42 (N=22;6;30) | 5 | 2 | 27
  LDH Above, Day 0 (N=22;6;29) | 18 | 4 | 3
  LDH Above, Day 7 (N=23;6;30) | 21 | 4 | 1
  LDH Above, Day 42 (N=22;6;30) | 16 | 4 | 3
  Sodium Unknown, Day 0 (N=22;6;29) | 0 | 0 | 0
  Sodium Unknown, Day 7 (N=23;6;30) | 0 | 0 | 0
  Sodium Unknown, Day 42 (N=22;6;30) | 0 | 0 | 0
  Sodium Below, Day 0 (N=22;6;29) | 0 | 0 | 0
  Sodium Below, Day 7 (N=23;6;30) | 0 | 0 | 0
  Sodium Below, Day 42 (N=22;6;30) | 0 | 0 | 0
  Sodium Within, Day 0 (N=22;6;29) | 22 | 6 | 29
  Sodium Within, Day 7 (N=23;6;30) | 23 | 6 | 30
  Sodium Within, Day 42 (N=22;6;30) | 22 | 6 | 30
  Sodium Above, Day 0 (N=22;6;29) | 0 | 0 | 0
  Sodium Above, Day 7 (N=23;6;30) | 0 | 0 | 0
  Sodium Above, Day 42 (N=22;6;30) | 0 | 0 | 0
  Protein Unknown, Day 0 (N=22;6;29) | 0 | 0 | 0
  Protein Unknown, Day 7 (N=23;6;30) | 0 | 0 | 0
  Protein Unknown, Day 42 (N=22;6;30) | 1 | 0 | 0
  Protein Below, Day 0 (N=22;6;29) | 2 | 0 | 4
  Protein Below, Day 7 (N=23;6;30) | 3 | 1 | 1
  Protein Below, Day 42 (N=22;6;30) | 2 | 0 | 3
  Protein Within, Day 0 (N=22;6;29) | 20 | 6 | 25
  Protein Within, Day 7 (N=23;6;30) | 20 | 5 | 29
  Protein Within, Day 42 (N=22;6;30) | 19 | 6 | 27
  Protein Above, Day 0 (N=22;6;29) | 0 | 0 | 0
  Protein Above, Day 7 (N=23;6;30) | 0 | 0 | 0
  Protein Above, Day 42 (N=22;6;30) | 0 | 0 | 0
  Urate/Uric acid Unknown, Day 0 (N=22;6;29) | 0 | 0 | 0
  Urate/Uric acid Unknown, Day 7 (N=23;6;30) | 0 | 0 | 0
  Urate/Uric acid Unknown, Day 42 (N=22;6;30) | 0 | 0 | 0
  Urate/Uric acid Below, Day 0 (N=22;6;29) | 9 | 2 | 0
  Urate/Uric acid Below, Day 7 (N=23;6;30) | 9 | 2 | 2
  Urate/Uric acid Below, Day 42 (N=22;6;30) | 9 | 2 | 2
  Urate/Uric acid Within, Day 0 (N=22;6;29) | 13 | 4 | 27
  Urate/Uric acid Within, Day 7 (N=23;6;30) | 14 | 4 | 26
  Urate/Uric acid Within, Day 42 (N=22;6;30) | 13 | 4 | 26
  Urate/Uric acid Above, Day 0 (N=22;6;29) | 0 | 0 | 2
  Urate/Uric acid Above, Day 7 (N=23;6;30) | 0 | 0 | 2
  Urate/Uric acid Above, Day 42 (N=22;6;30) | 0 | 0 | 2
  BUN Unknown, Day 0 (N=22;6;29) | 0 | 0 | 0
  BUN Unknown, Day 7 (N=23;6;30) | 0 | 0 | 0
  BUN Unknown, Day 42 (N=22;6;30) | 0 | 0 | 0
  BUN Below, Day 0 (N=22;6;29) | 0 | 0 | 0
  BUN Below, Day 7 (N=23;6;30) | 1 | 0 | 0
  BUN Below, Day 42 (N=22;6;30) | 0 | 0 | 1
  BUN Within, Day 0 (N=22;6;29) | 22 | 6 | 29
  BUN Within, Day 7 (N=23;6;30) | 21 | 6 | 30
  BUN Within, Day 42 (N=22;6;30) | 22 | 6 | 28
  BUN Above, Day 0 (N=22;6;29) | 0 | 0 | 0
  BUN Above, Day 7 (N=23;6;30) | 1 | 0 | 0
  BUN Above, Day 42 (N=22;6;30) | 0 | 0 | 1

38. Secondary Outcome: Number of Subjects With Normal or Abnormal Values of Haematological Parameters
Description: Among haematological parameters assessed were Basophils (Baso), Eosinophils (EOS), Hematocrit (HEM), Hemoglobin (Hgb), Lymphocytes (LYM), Monocytes (MON), Neutrophils (NEU), Platelets (PLA), Red Blood Cells (RBC) and White Blood Cells (WBC).
  Unknown = value unknown for the specified time point and laboratory parameter; Below = value below the laboratory reference range defined for the specified time point and laboratory parameter; Within = value within the laboratory reference range defined for the specified time point and laboratory parameter; Above = value above the laboratory reference range defined for the specified time point and laboratory parameter.
Time Frame: At Days 0, 7 and 42
Population: The analysis was performed on the Total Vaccinated Cohort, which included all vaccinated subjects.
Measure: Number; unit: Subjects
Arm/Group | GSK2340274A_F1 6M-5Y Subgroup | GSK2340274A_F1 6Y-9Y Subgroup | GSK2340274A_F2 10Y-17Y Group
Number analyzed (Participants) | 23 | 6 | 30
Subjects
  BAS Unknown, Day 0 (N=22;6;29) | 0 | 0 | 1
  BAS Unknown, Day 7 (N=23;6;30) | 0 | 0 | 0
  BAS Unknown, Day 42 (N=22;6;30) | 0 | 0 | 0
  BAS Below, Day 0 (N=22;6;29) | 0 | 0 | 0
  BAS Below, Day 7 (N=23;6;30) | 0 | 0 | 0
  BAS Below, Day 42 (N=22;6;30) | 0 | 0 | 0
  BAS Within, Day 0 (N=22;6;29) | 22 | 6 | 28
  BAS Within, Day 7 (N=23;6;30) | 23 | 6 | 30
  BAS Within, Day 42 (N=22;6;30) | 22 | 6 | 30
  BAS Above, Day 0 (N=22;6;29) | 0 | 0 | 0
  BAS Above, Day 7 (N=23;6;30) | 0 | 0 | 0
  BAS Above, Day 42 (N=22;6;30) | 0 | 0 | 0
  EOS Unknown, Day 0 (N=22;6;29) | 0 | 0 | 1
  EOS Unknown, Day 7 (N=23;6;30) | 0 | 0 | 0
  EOS Unknown, Day 42 (N=22;6;30) | 0 | 0 | 0
  EOS Below, Day 0 (N=22;6;29) | 0 | 0 | 0
  EOS Below, Day 7 (N=23;6;30) | 0 | 0 | 0
  EOS Below, Day 42 (N=22;6;30) | 0 | 0 | 0
  EOS Within, Day 0 (N=22;6;29) | 18 | 6 | 23
  EOS Within, Day 7 (N=23;6;30) | 21 | 6 | 25
  EOS Within, Day 42 (N=22;6;30) | 21 | 6 | 27
  EOS Above, Day 0 (N=22;6;29) | 4 | 0 | 5
  EOS Above, Day 7 (N=23;6;30) | 2 | 0 | 5
  EOS Above, Day 42 (N=22;6;30) | 1 | 0 | 3
  HEM Unknown, Day 0 (N=22;6;29) | 0 | 0 | 1
  HEM Unknown, Day 7 (N=23;6;30) | 0 | 0 | 0
  HEM Unknown, Day 42 (N=22;6;30) | 0 | 0 | 0
  HEM Below, Day 0 (N=22;6;29) | 7 | 3 | 1
  HEM Below, Day 7 (N=23;6;30) | 7 | 3 | 3
  HEM Below, Day 42 (N=22;6;30) | 9 | 3 | 4
  HEM Within, Day 0 (N=22;6;29) | 15 | 3 | 25
  HEM Within, Day 7 (N=23;6;30) | 16 | 3 | 26
  HEM Within, Day 42 (N=22;6;30) | 13 | 3 | 26
  HEM Above, Day 0 (N=22;6;29) | 0 | 0 | 2
  HEM Above, Day 7 (N=23;6;30) | 0 | 0 | 1
  HEM Above, Day 42 (N=22;6;30) | 0 | 0 | 0
  Hgb Unknown, Day 0 (N=22;6;29) | 0 | 0 | 1
  Hgb Unknown, Day 7 (N=23;6;30) | 0 | 0 | 0
  Hgb Unknown, Day 42 (N=22;6;30) | 0 | 0 | 0
  Hgb Below, Day 0 (N=22;6;29) | 10 | 3 | 8
  Hgb Below, Day 7 (N=23;6;30) | 10 | 4 | 8
  Hgb Below, Day 42 (N=22;6;30) | 12 | 3 | 6
  Hgb Within, Day 0 (N=22;6;29) | 12 | 3 | 20
  Hgb Within, Day 7 (N=23;6;30) | 13 | 2 | 22
  Hgb Within, Day 42 (N=22;6;30) | 10 | 3 | 24
  Hgb Above, Day 0 (N=22;6;29) | 0 | 0 | 0
  Hgb Above, Day 7 (N=23;6;30) | 0 | 0 | 0
  Hgb Above, Day 42 (N=22;6;30) | 0 | 0 | 0
  LYM Unknown, Day 0 (N=22;6;29) | 0 | 0 | 1
  LYM Unknown, Day 7 (N=23;6;30) | 0 | 0 | 0
  LYM Unknown, Day 42 (N=22;6;30) | 0 | 0 | 0
  LYM Below, Day 0 (N=22;6;29) | 0 | 0 | 0
  LYM Below, Day 7 (N=23;6;30) | 0 | 0 | 0
  LYM Below, Day 42 (N=22;6;30) | 0 | 0 | 0
  LYM Within, Day 0 (N=22;6;29) | 18 | 6 | 28
  LYM Within, Day 7 (N=23;6;30) | 17 | 6 | 29
  LYM Within, Day 42 (N=22;6;30) | 18 | 6 | 30
  LYM Above, Day 0 (N=22;6;29) | 4 | 0 | 0
  LYM Above, Day 7 (N=23;6;30) | 6 | 0 | 1
  LYM Above, Day 42 (N=22;6;30) | 4 | 0 | 0
  MON Unknown, Day 0 (N=22;6;29) | 0 | 0 | 1
  MON Unknown, Day 7 (N=23;6;30) | 0 | 0 | 0
  MON Unknown, Day 42 (N=22;6;30) | 0 | 0 | 0
  MON Below, Day 0 (N=22;6;29) | 0 | 0 | 0
  MON Below, Day 7 (N=23;6;30) | 0 | 0 | 0
  MON Below, Day 42 (N=22;6;30) | 0 | 0 | 0
  MON Within, Day 0 (N=22;6;29) | 21 | 6 | 27
  MON Within, Day 7 (N=23;6;30) | 21 | 6 | 29
  MON Within, Day 42 (N=22;6;30) | 22 | 6 | 28
  MON Above, Day 0 (N=22;6;29) | 1 | 0 | 1
  MON Above, Day 7 (N=23;6;30) | 2 | 0 | 1
  MON Above, Day 42 (N=22;6;30) | 0 | 0 | 2
  NEU Unknown, Day 0 (N=22;6;29) | 0 | 0 | 1
  NEU Unknown, Day 7 (N=23;6;30) | 0 | 0 | 0
  NEU Unknown, Day 42 (N=22;6;30) | 0 | 0 | 0
  NEU Below, Day 0 (N=22;6;29) | 8 | 0 | 1
  NEU Below, Day 7 (N=23;6;30) | 12 | 1 | 1
  NEU Below, Day 42 (N=22;6;30) | 7 | 0 | 1
  NEU Within, Day 0 (N=22;6;29) | 14 | 6 | 27
  NEU Within, Day 7 (N=23;6;30) | 11 | 5 | 29
  NEU Within, Day 42 (N=22;6;30) | 15 | 6 | 29
  NEU Above, Day 0 (N=22;6;29) | 0 | 0 | 0
  NEU Above, Day 7 (N=23;6;30) | 0 | 0 | 0
  NEU Above, Day 42 (N=22;6;30) | 0 | 0 | 0
  PLA Unknown, Day 0 (N=22;6;29) | 0 | 0 | 1
  PLA Unknown, Day 7 (N=23;6;30) | 0 | 0 | 0
  PLA Unknown, Day 42 (N=22;6;30) | 0 | 0 | 0
  PLA Below, Day 0 (N=22;6;29) | 1 | 0 | 0
  PLA Below, Day 7 (N=23;6;30) | 0 | 0 | 0
  PLA Below, Day 42 (N=22;6;30) | 1 | 0 | 0
  PLA Within, Day 0 (N=22;6;29) | 16 | 6 | 27
  PLA Within, Day 7 (N=23;6;30) | 14 | 5 | 29
  PLA Within, Day 42 (N=22;6;30) | 13 | 5 | 29
  PLA Above, Day 0 (N=22;6;29) | 5 | 0 | 1
  PLA Above, Day 7 (N=23;6;30) | 9 | 1 | 1
  PLA Above, Day 42 (N=22;6;30) | 8 | 1 | 1
  RBC Unknown, Day 0 (N=22;6;29) | 0 | 0 | 1
  RBC Unknown, Day 7 (N=23;6;30) | 0 | 0 | 0
  RBC Unknown, Day 42 (N=22;6;30) | 0 | 0 | 0
  RBC Below, Day 0 (N=22;6;29) | 0 | 0 | 0
  RBC Below, Day 7 (N=23;6;30) | 0 | 0 | 0
  RBC Below, Day 42 (N=22;6;30) | 0 | 1 | 0
  RBC Within, Day 0 (N=22;6;29) | 21 | 6 | 26
  RBC Within, Day 7 (N=23;6;30) | 22 | 6 | 28
  RBC Within, Day 42 (N=22;6;30) | 20 | 5 | 29
  RBC Above, Day 0 (N=22;6;29) | 1 | 0 | 2
  RBC Above, Day 7 (N=23;6;30) | 1 | 0 | 2
  RBC Above, Day 42 (N=22;6;30) | 2 | 0 | 1
  WBC Unknown, Day 0 (N=22;6;29) | 0 | 0 | 1
  WBC Unknown, Day 7 (N=23;6;30) | 0 | 0 | 0
  WBC Unknown, Day 42 (N=22;6;30) | 0 | 0 | 0
  WBC Below, Day 0 (N=22;6;29) | 0 | 0 | 0
  WBC Below, Day 7 (N=23;6;30) | 0 | 0 | 0
  WBC Below, Day 42 (N=22;6;30) | 0 | 0 | 0
  WBC Within, Day 0 (N=22;6;29) | 14 | 6 | 28
  WBC Within, Day 7 (N=23;6;30) | 10 | 5 | 30
  WBC Within, Day 42 (N=22;6;30) | 12 | 4 | 29
  WBC Above, Day 0 (N=22;6;29) | 8 | 0 | 0
  WBC Above, Day 7 (N=23;6;30) | 13 | 1 | 0
  WBC Above, Day 42 (N=22;6;30) | 10 | 2 | 1

ADVERSE EVENTS:
Time Frame: Solicited local and general symptoms: during the 7-day (Day 0-6) post-vaccination period; Unsolicited AEs: up to 84 days (Days 0-83) after the first vaccination; SAEs: during the entire study period (from Day 0 up to Day 182).
Arm/Group | GSK2340274A_F1 6M-9Y Group | GSK2340274A_F2 10Y-17Y Group
Serious Adverse Events (participants affected / at risk) | 1/30 | 1/30
Other Adverse Events (participants affected / at risk) | 30/30 | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GSK2340274A_F1 6M-9Y Group (N=30) | GSK2340274A_F2 10Y-17Y Group (N=30)
Febrile convulsion (Nervous system disorders) | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | GSK2340274A_F1 6M-9Y Group (N=30) | GSK2340274A_F2 10Y-17Y Group (N=30)
Pain (General disorders) | 25 | 30
Redness (General disorders) | 3 | 10
Swelling (General disorders) | 10 | 16
Drowsiness (6m-5y) (General disorders) | 8/24 | 0/0
Irritability (6m-5y) (General disorders) | 8/24 | 0/0
Loss of appetite (6m-5y) (General disorders) | 7/24 | 0/0
Fatigue (6y-9y + 10y-17y) (General disorders) | 2/6 | 14
Gastrointestinal (6y-9y + 10y-17y) (General disorders) | 2/6 | 4
Headache (6y-9y + 10y-17y) (General disorders) | 3/6 | 20
Joint pain (6y-9y + 10y-17y) (General disorders) | 0/6 | 9
Muscle aches (6y-9y + 10y-17y) (General disorders) | 0/6 | 11
Shivering (6y-9y + 10y-17y) (General disorders) | 1/6 | 11
Sweating (6y-9y + 10y-17y) (General disorders) | 0/6 | 5
Temperature (Axillary) (General disorders) | 10 | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 2
Pyrexia (General disorders) | 6 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 7 | 1
Upper respiratory tract infection (Infections and infestations) | 6 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 0
Gastroenteritis (Infections and infestations) | 3 | 0
Nasopharyngitis (Infections and infestations) | 3 | 1
Vomiting (Gastrointestinal disorders) | 3 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 2
Axillary pain (General disorders) | 0 | 2
Bronchitis (Infections and infestations) | 2 | 1
Eye discharge (Eye disorders) | 2 | 0
Headache (Nervous system disorders) | 0 | 2
Influenza (Infections and infestations) | 1 | 2
Pharyngitis (Infections and infestations) | 0 | 2
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.